CLINICAL TRIAL: NCT05089708
Title: Evaluation of Acne-induced Hyperpigmentation During Treatment of Acne Vulgaris Subjects With Trifarotene 50 μg/g Cream Versus Vehicle Cream Over 24 Weeks
Brief Title: AkLief Evaluation in Acne-induced Post-Inflammatory Hyperpigmentation
Acronym: LEAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.204245; 2021-003608-41 (EudraCT Number)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Trifarotene; Aklief; CD5789
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trifarotene (CD5789) 50 mcg/g Cream (Experimental)
  Interventions: Drug: Trifarotene Cream
- Trifarotene Vehicle Cream (Placebo Comparator)
  Interventions: Drug: Trifarotene Vehicle Cream

INTERVENTIONS:
Drug: Trifarotene Cream — Participants will apply a thin a layer of trifarotene (CD5789) 50 mcg/g cream on the face once daily, in the evening for 24 weeks
  Other Names: Aklief
  Arms: Trifarotene (CD5789) 50 mcg/g Cream
Drug: Trifarotene Vehicle Cream — Participants will apply a thin a layer of trifarotene vehicle cream on the face once daily, in the evening for 24 weeks
  Arms: Trifarotene Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Trifarotene 50 microgram per gram (mcg/g) cream compared to its vehicle cream in the treatment of moderate acne vulgaris with risk of acne-induced post inflammatory hyperpigmentation (PIH) after 24 weeks of treatment in facial acne participants

ELIGIBILITY:
Key Inclusion Criteria:

* Participant with clinical diagnosis of acne vulgaris, defined by:

  1. moderate acne on the face (acne Investigator's Global Assessment [IGA] =3); and
  2. with minimum of 20 inflammatory lesions and 25 non inflammatory lesions on the face (excluding the nose); and
  3. moderate to marked PIH on the face (Overview of Pigmentation Disorders hyperpigmentation scale 4-6); and
  4. no more than one acne nodule or cyst (greater than [>] 1 centimeter [cm]) on face (excluding the nose)
* Participant with any Fitzpatrick Skin Type I to VI (target patient enrollment according to FST)
* Female participants of childbearing potential must have a negative urine pregnancy test (UPT) at Baseline visit
* Female participants of childbearing potential must agree to use an adequate and approved method of contraception throughout the study
* Female participant of non-childbearing potential
* Other protocol defined inclusion criteria could apply

Key Exclusion Criteria:

* Participant with severe acne (IGA > 3)
* Participant with more than 1 nodule/cyst on the face (excluding the nose)
* Participant with acne conglobata, acne fulminans, secondary acne, nodulocystic acne, acne requiring systemic treatment
* Participant with damaged facial skin that may interfere with study assessments
* Female participant who is pregnant, lactating or planning a pregnancy during the study
* Female participant of childbearing potential using combined oral contraceptives approved as acne treatments, in whom the dose has not been stable for at least 6 months prior to the Baseline visit
* Participant with known impaired hepatic or renal functions
* Participant with active or chronic skin allergies

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (22):
  - Galderma Investigational Site #8636, Fountain Valley, California
  - Galderma Investigational Site #8224, Fremont, California
  - Galderma Investigational Site #8358, San Diego, California
  - Galderma Investigational Site #9955, San Diego, California
  - Galderma Investigational Site #7012, Lutz, Florida
  - Galderma Investigational Site #8184, Maitland, Florida
  - Galderma Investigational Site #8764, Tampa, Florida
  - Galderma Investigational Site #9950, Evansville, Indiana
  - Galderma Investigational Site #9952, Baton Rouge, Louisiana
  - Galderma Investigational Site #8606, New Orleans, Louisiana
  - Galderma Investigational Site #8012, Glenn Dale, Maryland
  - Galderma Investigational Site #9948, Hyattsville, Maryland
  - Galderma Investigational Site #8554, Detroit, Michigan
  - Galderma Investigational Site #8108, Las Vegas, Nevada
  - Galderma Investigational Site #8620, New York, New York
  - Galderma Investigational Site #9956, New York, New York
  - Galderma Investigational Site #9949, New York, New York
  - Galderma Investigational Site #9953, Tulsa, Oklahoma
  - Galderma Investigational Site #8207, Nashville, Tennessee
  - Galderma Investigational Site #9920, Arlington, Texas
  - Galderma Investigational Site #8329, San Antonio, Texas
  - Galderma Investigational Site #8433, San Antonio, Texas
- Spain (3):
  - Galderma Investigational Site #6192, Zaragoza, Aragon
  - Galderma Investigational Site #6278, Manises, Valencia
  - Galderma Investigational Site #6277, Pontevedra

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 investigational centers in the United States and Spain from 22 Dec 2021 to 15 Dec 2022.
Pre-assignment Details: A total of 150 participants were screened, out of which 123 participants were randomized and enrolled in two treatment groups. 60 participants were randomized in Trifarotene (CD5789) Cream treatment group and 63 were assigned in Trifarotene Vehicle Cream treatment group.
Groups:
- Trifarotene (CD5789) Cream: Participants applied Trifarotene 50 micrograms per gram (mcg/g) cream on face once daily in the evening for 24 weeks.
- Trifarotene Vehicle Cream: Participants applied Trifarotene Vehicle cream on face once daily in the evening for 24 weeks.
Period: Overall Study
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream
Started | 60 | 63
Completed | 45 | 53
Not Completed | 15 | 10
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Non-Compliance with Investigational Product | 1 | 1
Not completed — Withdrawal by Parent or Guardian | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Trifarotene (CD5789) Cream: Participants applied Trifarotene 50 mcg/g cream on face once daily in the evening for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (6.30) | 21.9 (5.95) | 22.3 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 93
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 27 | 48
  Not Hispanic or Latino | 39 | 36 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 22 | 23 | 45
  White | 25 | 31 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Post-Inflammatory Hyperpigmentation (PIH) Overall Disease Severity (ODS) Scores at Week 24
Description: The PIH ODS Score is based on a 9-point scale: Grade 0 Normal; Grade 1 Present, but <mild; Grade 2 Mild (slightly noticeable); Grade 3 Between mild and moderate; Grade 4 Moderate; Grade 5 Between moderate and marked; Grade 6 Marked (distinctive); Grade 7 Between marked and severe; Grade 8 Severe (very distinctive). A negative change indicates a reduction from in PIH disease severity score from baseline.
Time Frame: Baseline and Week 24
Population: The Intent to Treat (ITT) population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream
Number analyzed (Participants) | 60 | 63
score on a scale | -2.1 (0.27) | -2.1 (0.24)

2. Secondary Outcome: Percent Change From Baseline in PIH ODS Scores at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream
Number analyzed (Participants) | 60 | 63
Percent change | -45.4 (5.73) | -44.9 (5.18)

3. Secondary Outcome: Absolute Change From Baseline in PIH ODS Scores at Weeks 12, 16 and 20
Description: as for outcome 1
Time Frame: Baseline, at Week 12, Week 16 and Week 20
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Trifarotene (CD5789) Cream: Participants applied Trifarotene 50 mcg/g cream on face once daily for 24 weeks.
- Trifarotene Vehicle Cream: Participants applied Trifarotene Vehicle cream on face once daily for 24 weeks.
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream
Number analyzed (Participants) | 60 | 63
score on a scale
  Absolute change at Week 12 | -1.6 (0.18) | -1.1 (0.17)
  Absolute change at Week 16 | -1.9 (0.2) | -1.7 (0.19)
  Absolute change at Week 20 | -2.0 (0.22) | -1.9 (0.21)

4. Secondary Outcome: Percent Change From Baseline in PIH Overall Disease Severity Scores at Weeks 12, 16 and 20
Description: as for outcome 1
Time Frame: Baseline, at Week 12, Week 16 and Week 20
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream
Number analyzed (Participants) | 60 | 63
Percent change
  Percent Change at Week 12 | -34.4 (3.78) | -23.6 (3.60)
  Percent Change at Week 16 | -41.2 (4.35) | -36.1 (4.17)
  Percent Change at Week 20 | -43.9 (4.83) | -41.0 (4.75)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from screening up to Week 24
Arm/Group | Trifarotene (CD5789) Cream | Trifarotene Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/63
Other Adverse Events (participants affected / at risk) | 10/60 | 19/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifarotene (CD5789) Cream (N=60) | Trifarotene Vehicle Cream (N=63)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifarotene (CD5789) Cream (N=60) | Trifarotene Vehicle Cream (N=63)
COVID-19 (Infections and infestations) | 3 (3) | 6 (6)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headached (Nervous system disorders) | 0 (0) | 2 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Application site burn (General disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT05089708/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT05089708/SAP_001.pdf